CLINICAL TRIAL: NCT02913274
Title: Fistules Artério-Veineuses: Angioplastie Par Ballon à Elution de Drogue (FAVABED) - Arteriovenous Fistulae: Drug-eluting Balloon Angioplasty
Brief Title: Arteriovenous Fistulae: Drug-eluting Balloon Angioplasty
Acronym: FAVABED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was temporarily suspended after a meta-analysis suggesting higher mortality risks among patients treated with Paclitaxel-coated balloons. When the study was open again, no new patient accepted to be included. The study stopped on 18AUG2023.
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-A00420-51
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "DEB" arm (Experimental): dilation by a high-pressure conventional angioplasty balloon (sized to fit the reference native vein diameter) until disappearance of the stenotic obstructive area and achievement of technical success (possibility of changing balloon size or dilation pressure) then dilation by a DEB.
  Interventions: Device: Paclitaxel (Taxol) eluting angioplasty balloon; Device: high-pressure angioplasty balloon
- "conventional angioplasty" arm (Active Comparator): dilation will be performed by a conventional high-pressure balloon until technical success is achieved (possibility of changing balloon size or dilation pressure), then by a sham balloon i.e a conventional low-pressure balloon (placebo)
  Interventions: Device: high-pressure angioplasty balloon; Device: low-pressure balloon

INTERVENTIONS:
Device: Paclitaxel (Taxol) eluting angioplasty balloon — Dilatation by a high-pressure conventional angioplasty balloon untill disappearance of the stenosis obstructive area and achievement of technical success. Then dilatation by a DEB of the same size for 2 minutes.
  Other Names: BARD, Lutonix® 035 and Lutonix®5F GeoAlign™
  Arms: "DEB" arm
Device: high-pressure angioplasty balloon — Dilatation by a high-pressure conventional angioplasty balloon untill disappearance of the stenosis obstructive area and achievement of technical success. Then dilatation either by a shame balloon or by a DEB balloon of the same size for 2 minutes.
  Other Names: BARD, Conquest®
Device: low-pressure balloon — Dilatation by a high-pressure conventional angioplasty balloon untill disappearance of the stenosis obstructive area and achievement of technical success. Thenn dilatation by a shame balloon i.e conventional low pression balloon of the same size for 2 minutes.
  Other Names: BARD, Ultraverse®
  Arms: "conventional angioplasty" arm

SUMMARY:
Dysfunctions such as tight stenosis or thrombosis in haemodialysis vascular accesses are the leading cause of hospitalisationand morbidity in chronic haemodialysis patients incurring significant related costs estimated at over one billion dollars in the USA.

Dysfunctions of these vascular accesses are generally treated by conventional angioplasty as this is the least invasive procedure, the alternative being revision surgery. Angioplasty uses an inflatable balloon of various diameters. Different types of angioplasty balloons may be needed to break fibrous venous stenosis, in particular high-pressure balloons or cutting balloons. These angioplasty procedures which are often painful during dilation have a high technical success rate but a poor 1-year patency rate.

These invasive repeated procedures impair the quality of life of these patients with end-stage renal disease who are on permanent dialysis or awaiting a kidney transplant and for whom vascular access patency is vital.

Due to their traumatic effect on the vessel wall, these procedures induce cell proliferation processes that retrigger neointimal hyperplasia the very act of preserving the haemodialysis access is the key factor in development of a new stenosis and hence a vicious circle of stenosis-angioplasty.

For the past few years, angioplasty balloons delivering anticancer drugs have been developed. These drugs, generally used in high doses for cancer chemotherapy, are released in small doses on the medical angioplasty devices. During inflation, the local release of the anticancer molecule through the different layers of the vessel wall confers local antiproliferative action without the systemic toxic effects associated with high-dose chemotherapy.

These medical devices have demonstrated their efficacy in terms of increase in primary and secondary patency rates on procedures such as coronary artery angioplasty, femoro-popliteal or sub-popliteal artery angioplasty.

These drug-eluting balloons (DEBs) are also CE marked with the recommendation of being indicated for AVF anticancerangioplasties, but no randomised multi-centre clinical trial has proven their medical effectiveness, and in particular their contribution in terms of patency rate improvement. However, studies on animal models show significant results regarding efficacy against neointimal hyperplasia and the first single-centre clinical trials on a small sample size appear promising.

The key assessment criterion is primary patency of the dilated stenosis at one year defined by patients efficaciously dialysed at one year without re-intervention on the dilated lesion after initial angioplasty. The delay of occurrence of dilation will be considered. Patients that will be non-evaluable for the primary endpointwill be censored at the date of the latest news.

DETAILED DESCRIPTION:
Dysfunctions such as tight stenosis or thrombosis in haemodialysis vascular accesses are the leading cause of hospitalisation (20%) and morbidity in chronic haemodialysis patients incurring significant related costs estimated at over one billion dollars in the USA.

Dysfunctions of these vascular accesses are generally treated by conventional angioplasty as this is the least invasive procedure, the alternative being revision surgery. Angioplasty uses an inflatable balloon of various diameters. Different types of angioplasty balloons may be needed to break fibrous venous stenosis, in particular high-pressure balloons (20 atm) or cutting balloons. These angioplasty procedures which are often painful during dilation have a high technical success rate (90-97%) but a poor 1-year patency rate, varying between 26 and 64% depending on the team and a mean rate estimated at 40% for the studies including the larger number of patients, some of whom requiring several procedures.

These invasive repeated procedures impair the quality of life of these patients with end-stage renal disease who are on permanent dialysis or awaiting a kidney transplant and for whom vascular access patency is vital.

Due to their traumatic effect on the vessel wall, these procedures induce cell proliferation processes that retrigger neointimal hyperplasia the very act of preserving the haemodialysis access is the key factor in development of a new stenosis and hence a vicious circle of stenosis-angioplasty.

For the past few years, angioplasty balloons delivering anticancer drugs (Paclitaxel, Sirolimus, Everolimus) have been developed. These drugs, generally used in high doses for cancer chemotherapy, are released in small doses on the medical angioplasty devices. During inflation, the local release of the anticancer (antimitotic) molecule through the different layers of the vessel wall (Paclitaxel is lipophilic and hydrophobic) confers local antiproliferative action without the systemic toxic effects associated with high-dose chemotherapy.

These medical devices have demonstrated their efficacy in terms of increase in primary and secondary patency rates on procedures such as coronary artery angioplasty, femoro-popliteal or sub-popliteal artery angioplasty (treatment of angina or lower limb arteriopathy).

These drug-eluting balloons (DEBs) are also CE marked with the recommendation of being indicated for AVF anticancerangioplasties, but no randomised multi-centre clinical trial has proven their medical effectiveness, and in particular their contribution in terms of patency rate improvement. However, studies on animal models show significant results regarding efficacy against neointimal hyperplasia and the first single-centre clinical trials on a small sample size appear promising.

The key assessment criterion is primary patency of the dilated stenosis at one year defined by patients efficaciously dialysed at one year without re-intervention on the dilated lesion after initial angioplasty. The delay of occurrence of dilation will be considered (censored criteria). Patients that will be non-evaluable for the primary endpoint (death, lost to follow-up…) will be censored at the date of the latest news.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18,
* Stage 5 renal failure patients on permanent haemodialysis treatment (every 2 or 3 days),
* Native and efficient arteriovenous fistula > 3 months,
* 3mm ≤ reference vein diameter ≤ 8 mm and stenosis length ≤ 10 cm (range of DEB diameters and lengths),
* Absence of fistula thrombosis,
* Possibility of crossing the stenosis with a guide wire,
* Significant stenosis > 50% (in relation to the reference diameter) on the fistulogram,
* Clinical diagnosis of imminent fistula dysfunction

  * pressure rise during dialysis
  * and/or puncture difficulties
  * and/or recirculation or poor extrarenal clearance
  * and/or decrease in vascular access flow
  * and/or increase in compression time after dialysis
* Social security affiliation,
* Receipt of free, informed, written consent.

Exclusion Criteria:

* Multiple stenoses,
* Goretex® graft prostheses
* Systemic or local infection,
* Known allergy to contrast agent or Paclitaxel.
* Comorbidity not permitting long-term follow-up,
* Life expectancy < 1 year,
* Anticancer treatment (patients treated with chemotherapy for neoplasia),
* Pregnant or breastfeeding woman,
* Patients over 18 years of age who are under legal protection (conservatorship, trusteeship, guardianship), or deprived of freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Number of patients whose haemodialysis is efficient at 1 year without needing further treatment of the stenotic site after initial angioplasty | 1 year
  assess the primary patency at 1 year after the dilatation of native AVF stenosis with "active" drug-eluting balloons (DEB) compared to conventional "plain" balloons, i.e to compare between the two groups the number of patients whose haemodialysis is efficient at 1 year without needing further treatment of the stenotic site after initial angioplasty.

SECONDARY OUTCOMES:
primary patency at 6 months | 6 months
  assess the advantages of Drug-Eluting Balloon compared to conventional plain balloon for primary patency at 6 months of the dilated stenosis
overall primary patency of the Arteriovenous Fistula at 1 year | 1 year
  assess the advantages of Drug-Eluting Balloon compared to conventional plain balloon for overall primary patency of the Arteriovenous Fistula at 1 year (patency including AVF dysfunction in relation to the initial dilated stenosis as well as stenoses distant from the initially treated site)
assisted primary patency of the dilated stenosis at 1 year | 1 year
  assess the advantages of Drug-Eluting Balloon compared to conventional plain balloon for assisted primary patency of the dilated stenosis at 1 year: Arteriovenous Fistula patency and continuation of efficient haemodialysis sessions with new angioplasties on the initially dilated stenotic site (excluding de-obstruction for complete thrombosis)
secondary patency of the AVF at 1 year | 1 year
  assess the advantages of Drug-Eluting Balloon compared to conventional plain balloon for secondary patency of the Arteriovenous Fistula at 1 year: Arteriovenous Fistula patency and continuation of efficient haemodialysis sessions also including complete thrombosis de-obstruction procedures
The minimal diameter of the treated stenosis and the AVF flows | 1 year
  assess the advantages of Drug-Eluting Balloon compared to conventional plain balloon for the minimal diameter of the treated stenosis (Late Luminal Loss) and the Arteriovenous Fistula flows (both criterion being evaluated by Doppler ultrasound and Transonic® after angioplasty, and at 6 months and 1 year follow-up).
Overall and cardiovascular survival | 5 years
  during analysis in sub-groups, the advantage of these Drug-Eluting Balloons for Overall and cardiovascular survival at 2 and 5 years for all patients and for subgroup of patients with symptomatic peripheral artery disease

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Heautot, MD, Principal Investigator — Rennes University Hospital
Locations (10):
- France (10):
  - CHU Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier d'Haguenau, Haguenau
  - APHM Hôpital la Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire de RENNES, Rennes
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Clinique St Gatien de Tours, Tours